CLINICAL TRIAL: NCT03710239
Title: OPIOID Study: Opioid Use and Pain After Insertion of Osmotic Dilators
Brief Title: OPIOID Study - Pain With Osmotic Dilators
Acronym: OPIOID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5209
Record Dates: First submitted 2018-10-14; First posted 2018-10-18 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Abortion in Second Trimester

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive one of two existing dilator times, with the remainder of care and study procedures being identical.
Who Masked: Participant
Masking Description: Participants will not know what type of dilator they have been assigned, however the medical care team (including investigators) will be aware.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dilapan-S (Active Comparator): Synthetic osmotic dilator
  Interventions: Device: Dilapan-S
- Laminaria (Active Comparator): Seaweed-based osmotic dilator
  Interventions: Device: Laminaria

INTERVENTIONS:
Device: Dilapan-S — Synthetic osmotic dilator
  Arms: Dilapan-S
Device: Laminaria — Seaweed-based osmotic dilator
  Arms: Laminaria

SUMMARY:
Comparison of pain levels and pain medications utilized following insertion of two different types of osmotic dilators.

DETAILED DESCRIPTION:
This is a randomized controlled trial to assess and compare pain levels and pain medication needs following placement of Laminaria versus Dilapan-S for cervical preparation prior to second-trimester dilation and evacuation (D&E) procedures. Pain levels and medication usage will also be assessed following the D&E procedure itself, up to 7 days after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* scheduled D&E for 15+0 to 23+6 wga
* ability to speak and read in English
* ownership of smartphone with internet access and data plan

Exclusion Criteria:

- chronic pain, fibromyalgia, active pelvic infection, inability to take NSAIDS, current use of narcotics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Maximum pain above baseline following Laminaria versus Dilapan-S placement | First 24 hours after dilator placement
  Timed surveys measuring pain on Numeric Rating Scale (0-10), administered approximately 24 hours after dilator placement
Time of maximum pain above baseline following Laminaria versus Dilapan-S placement | First 24 hours after dilator placement
  Timing of maximum Numeric Rating Scale (0-10) pain difference among measurements approximately 24 hours after dilator placement

SECONDARY OUTCOMES:
Pain medication use after Laminaria versus Dilapan-S placement | First 24 hours after dilator placement
  Timed surveys of pain medication usage at 2 hours, 4 hours, 8 hours, and approximately 24 hours after dilator placement
Maximum pain increase over baseline following D&E procedure | First week after D&E
  Timed surveys measuring pain on Numeric Rating Scale (0-10), administered at 1 hour, 4 hours, 24 hours, 48 hours, and 1 week after D&E procedure
Pain medication use after D&E | First week after D&E
  Timed surveys of pain medication usage, administered at 4 hours, 24 hours, 48 hours, and 1 week after D&E procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center Obstetrics and Gynecology, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No